CLINICAL TRIAL: NCT06191627
Title: Legs vs Back: Patient Experience and Quality of Patch Testing for Allergic Contact Dermatitis on Different Body Sites
Brief Title: Patient Experience and Quality of Patch Testing on the Legs vs Back
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A23-305
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2023-12

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Intervention Model Description: This study is a two-armed randomized trial. Patients will be recruited from the cohort already undergoing patch testing at our clinic. Enrolled and consented patients will be randomized in a 1:1 ratio to the legs or back study arm via a predetermined randomization order. Patches will be placed as indicated per each patient case, either on the thighs or back. At the 48-hr time point, patches will be removed. Study coordinators will grade success of testing by noting total patches applied and counting patches with a complete circular indentation, partial indentation, or absent indentation from the Finn chambers. Patients will then complete a survey prior to interpretation of their testing by the physician. The predetermined randomization order and survey data will be stored in the secure PN server.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patch testing on the legs (Active Comparator): Patches to be applied on the legs
  Interventions: Diagnostic Test: Patch testing
- Patch testing on the back (Active Comparator): Patches to be applied on the back
  Interventions: Diagnostic Test: Patch testing

INTERVENTIONS:
Diagnostic Test: Patch testing — Unlike many different dermatological diseases, a biopsy cannot easily distinguish ACD from irritant contact dermatitis or other forms of chronic dermatitis. Thus, the gold standard for diagnosis is patch testing. During patch testing, allergens are placed on the skin under occlusion using an aluminum disc and tape. When undergoing intensive testing for ACD, as many as 300 patches may be applied to a patient. Therefore, a large area of skin clear of rash is required, most often the back, but patches are frequently applied to the legs as well. Patches are applied by clinic patch technicians. They will proceed with their normal procedures, following the randomization to apply the patches to the appropriate location. Patches will be applied to the skin once, as is the normal standard of care. Patches are applied on day 1 and removed on day 3. Patients continue testing through day 5, though study elements will cease on day 3.

SUMMARY:
The gold standard for the diagnosis of allergic contact dermatitis is patch testing, during which allergens are affixed to the skin underneath tape and left for multiple days. A large area of clear skin is thus required for successful testing.

While the back is traditionally thought to be the ideal area for testing, the thighs may be more available or advantageous. This study seeks to randomize patients undergoing patch testing to have patches placed on the back or the thighs. The investigators seek to understand the benefits of testing on the legs versus the back in terms of patient experience as well as achieving a successful test. This study will measure patient experience using a survey administered to patients. Quality of testing will be assessed by study coordinators prior the removal of patches.

DETAILED DESCRIPTION:
Background:

Patch testing for ACD is a rigorous process. While the patches are on the patient's skin, they must be careful not to perform movements that will cause the tape to detach, thus compromising the integrity of the test. The classical placement of patches is on the back due to: a) the large body surface area in which to place the patches, b) the generally flat surface which allows for adequate adhesion of the patches (as opposed to a more rounded body surface), and c) the difficulty for patients to manipulate the area, thus limiting patient interference with the testing site and ensuring the tape remains adhered. The primary disadvantages of placing patches on one's back are the physical limitations, e.g the inability to raise one's arms above shoulder level, bend, twist, or reach. This has both comfort and practical disadvantages as patients find it hard to drive, clothe, and perform their activities of daily living (ADLs). These limitations improve the quality of the testing, but it is reasonable to think that some discomfort could be prevented, as an element of the physical limitations result from pulling or tugging due to the copious amounts of tape applied to achieve complete occlusion. For patients who are parents or caregivers, or those who are unable to take off of work during the week, these limitations can prove to be an immense challenge. Breastfeeding mothers may be unable to comfortably feed their infants. Patients also report increased pain, sleeping difficulties, and worsening of rash during patch testing.

Thus, the investigators seek to investigate further patient comfort during patch testing to improve the patient experience. The thighs have been used in our clinic as a patch testing as an alternative to the back, either when the back has rash, tattoos, or too small an area for complete patch testing. Anecdotal evidence suggests that the thighs may provide a more pleasant patch testing experience with decreased restrictions in mobility. In our experience, no limitation has been seen in terms of the quality of the patches with placement on the thighs. To date, there has been little published literature regarding the ideal location of patch testing, either in respect to patient experience or quality of testing. One study has proposed alternatives to the tape used to adhere patches in an effort to improve comfort. Another study examined retrospective data to identify rates of symptoms during patch testing (pain, sleep difficulty, need for medication, site itching or itching elsewhere, and worsening rash) and their correlation with patch location. Various significant statistical associations were found, such as highest levels of pain with placement on the arms and increased need for medication and location on the chest. However, more information is needed comparing specifically the legs and the back, the two most commonly tested areas, in terms of patient comfort and quality of the test. Additionally, by obtaining a more holistic understanding of patient comfort, the investigators will be able to derive a more useful and clinically applicable answer as to whether the legs or back is preferable for testing location.

Sample Size:

Sample size will be determined using a pragmatic approach based on time constraints and size of recruitment pool. Because there exists no previously validated instrument to measure patient experience during patch testing (or something similar), the investigators will be developing our own survey. The survey will document important demographic information and assess patient experience during patch testing using agreements questions that will be compared between both groups. HealthPartners Center for Evaluation and Survey Research (CESR) will help to develop an effective instrument. 30 patients will be enrolled per treatment group. Between 10-20 patients are seen per week on average, and the investigators estimate that 20% will not meet inclusion criteria. Assuming that 50% of patients who meet enrollment criteria will agree to take part in the study, data collection will take between 8-15 weeks. 100% study follow through should be attainable, as it is very rare for patients who begin patch testing to be lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergoing patch testing at Park Nicollet Contact Dermatitis
* At least 90 patches applied at one time, representing comprehensive testing rather than limited testing with few patches that may skew results
* Both back and thighs adequate for patch testing (see exclusion criteria below)

Exclusion Criteria:

* Patient is 17 or younger
* Patient is pregnant or breastfeeding
* Specialized patch testing with low number of patches (less than 90)
* Rash that would preclude testing on thighs or back
* Large tattoos that would preclude testing on thighs or back
* Limited space on thighs or back due to body habitus
* Patient has specific needs necessitating use of the thighs or back (event, breastfeeding, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Comfort during patch testing | Survey completed on day 3 of testing, taking no more than 10 minutes to complete.
  Patients in both arms will complete a survey that assesses their comfort while wearing patches as part of patch testing. The survey will be the same for both arms of the study. The primary outcome will consist of level of agreement with statements.
Quality of patch testing | Study coordinators will document the percentage of patches with appropriate occlusion on day 3 of testing prior to survey completion.
  The quality of patch testing in both arms will also be assessed. This will be based on the percentage of patches with appropriate occlusion. This will be defined by the presence of indentation made by the aluminum discs used for patching.

SECONDARY OUTCOMES:
Qualitative Survey Feedback | Survey collected on day 5
  Participants in both study arms will be able to leave qualitative feedback at the end of their survey. Any qualitative feedback left will be compared between both study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hylwa, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Contact Dermatitis Clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nassau S, Fonacier L. Allergic Contact Dermatitis. Med Clin North Am. 2020 Jan;104(1):61-76. doi: 10.1016/j.mcna.2019.08.012. Epub 2019 Oct 28. PMID 31757238
- [Result] Wildemore JK, Junkins-Hopkins JM, James WD. Evaluation of the histologic characteristics of patch test confirmed allergic contact dermatitis. J Am Acad Dermatol. 2003 Aug;49(2):243-8. doi: 10.1067/s0190-9622(03)00865-x. PMID 12894072
- [Result] Burkemper NM. Contact Dermatitis, Patch Testing, and Allergen Avoidance. Mo Med. 2015 Jul-Aug;112(4):296-300. PMID 26455061
- [Result] Kimyon RS, Hylwa SA, Neeley AB, Warshaw EM. Patch Testing: The Patient Experience. Dermatitis. 2021 Sep-Oct 01;32(5):333-338. doi: 10.1097/DER.0000000000000656. PMID 33273240
- [Result] Rodriguez-Lomba E, Sanchez-Herrero A, Morales P, Suarez-Fernandez R. Transparent Film Dressings for Patch Testing Leads to Better Adhesion and Patient Comfort. Dermatitis. 2018 Sep/Oct;29(5):289. doi: 10.1097/DER.0000000000000398. No abstract available. PMID 30179972

DOCUMENTS (1):
  • Informed Consent Form (2023-12-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT06191627/ICF_000.pdf